CLINICAL TRIAL: NCT04630808
Title: A Phase 3, Randomized, Multi-Regional, Double-Masked, Parallel-Group Trial Evaluating the Safety and Efficacy of NCX 470 0.1% vs. Latanoprost 0.005% in Subjects With Open-Angle Glaucoma or Ocular Hypertension (Denali)
Brief Title: MRCT Evaluating NCX 470 vs. Latanoprost in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Acronym: Denali
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nicox Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCX-470-03
Record Dates: First submitted 2020-11-11; First posted 2020-11-16 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NCX 470 0.1% (Experimental): NCX 470 Ophthalmic Solution, 0.1% dosed once daily to both eyes
  Interventions: Drug: NCX 470 0.1%
- Latanoprost 0.005% (Active Comparator): Latanoprost Ophthalmic Solution, 0.005% dosed once daily to both eyes
  Interventions: Drug: Latanoprost 0.005%

INTERVENTIONS:
Drug: NCX 470 0.1% — NCX 470 Ophthalmic Solution, 0.1%
  Other Names: NCX 470
  Arms: NCX 470 0.1%
Drug: Latanoprost 0.005% — Latanoprost Ophthalmic Solution, 0.005%
  Other Names: Latanoprost
  Arms: Latanoprost 0.005%

SUMMARY:
The objective of this clinical study is to evaluate the safety and efficacy of NCX 470 Ophthalmic Solution in lowering intraocular pressure (IOP) in subjecs with ocular hypertension or open-angle glaucoma. Subjects will be randomized in a 1:1 ratio to NCX 470 0.1% or to latanoprost 0.005% to be administered to both eyes once daily in the evening for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma or ocular hypertension in both eyes
* Qualifying IOP at 3 time points through the day at 2 visits following washout of IOP-lowering medication, if applicable
* Qualifying best-corrected visual acuity in each eye
* Ability to provide informed consent and follow study instructions

Exclusion Criteria:

* Narrow anterior chamber angles or disqualifying corneal thickness in either eye
* Clinically significant ocular disease in either eye
* Previous complicated surgery or certain types of glaucoma surgery in either eye
* Incisional ocular surgery or severe trauma in either eye within the past 6 months
* Uncontrolled systemic disease

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline IOP | Up to 3 months
  Mean IOP change from time-matched baseline at 8AM and 4PM time points at the Week 2, Week 6 and Month 3 Visits in the study eye

SECONDARY OUTCOMES:
Change from baseline in diurnal IOP | Up to 3 months
  Mean diurnal IOP change from baseline at the Week 2, Week 6 and Month 3 Visits in the study eye
Frequency and incidence of treatment-emergent adverse events | 12 months
  Number and percentage of subjects with ocular and non-ocular treatment-emergent adverse events
Rate of discontinuation | 12 months
  Percentage of subjects in each treatment group who discontinue study participation

CONTACTS AND LOCATIONS:
Overall Officials: Nicox Ophthalmics, Study Director — Nicox Ophthalmics, Inc.
Locations (77):
- United States (57):
  - Nicox Clinical Site, Dothan, Alabama
  - Nicox Clinical Site, Chandler, Arizona
  - Nicox Clinical Site, Phoenix, Arizona
  - Nicox Clinical Site, Burbank, California
  - Nicox Clinical Site, Garden Grove, California
  - Nicox Clinical Site, Huntington Beach, California
  - Nicox Clinical Site, La Jolla, California
  - Nicox Clinical Site, Murrieta, California
  - Nicox Clinical Site, Newport Beach, California
  - Nicox Clinical Site, Pasadena, California
  - Nicox Clinical Site, Petaluma, California
  - Nicox Clinical Site, Redlands, California
  - Nicox Clinical Site, San Francisco, California
  - Nicox Clinical Site, Danbury, Connecticut
  - Nicox Clinical Site, Boynton Beach, Florida
  - Nicox Clinical Site, Delray Beach, Florida
  - Nicox Clinical Site, Fort Lauderdale, Florida
  - Nicox Clinical Site, Fort Myers, Florida
  - Nicox Clinical Site, Jacksonville, Florida
  - Nicox Clinical Site, Jupiter, Florida
  - Nicox Clinical Site, Lakeland, Florida
  - Nicox Clinical Site, Largo, Florida
  - Nicox Clinical Site, Mt. Dora, Florida
  - Nicox Clinical Site, Venice, Florida
  - Nicox Clinical Site, Morrow, Georgia
  - Nicox Clinical Site, Roswell, Georgia
  - Nicox Clinical Site, Peoria, Illinois
  - Nicox Clinical Site, Rock Island, Illinois
  - Nicox Clinical Site, Indianapolis, Indiana
  - Nicox Clinical Site, Bangor, Maine
  - Nicox Clinical Site, Boston, Massachusetts
  - Nicox Clinical Site, Lancaster, Massachusetts
  - Nicox Clinical Site, Grand Rapids, Michigan
  - Nicox Clinical Site, Chaska, Minnesota
  - Nicox Clinical Site, Kansas City, Missouri
  - Nicox Clinical Site, St Louis, Missouri
  - Nicox Clinical Site, Clifton Park, New York
  - Nicox Clinical Site, The Bronx, New York
  - Nicox Clinical Site, Troy, New York
  - Nicox Clinical Site, Asheville, North Carolina
  - Nicox Clinical Site, Winston-Salem, North Carolina
  - Nicox Clinical Site, Fargo, North Dakota
  - Nicox Clinical Site, Cincinnati, Ohio
  - Nicox Clinical Site, Eugene, Oregon
  - Nicox Clinical Site, Cranberry Township, Pennsylvania
  - Nicox Clinical Site, Kingston, Pennsylvania
  - Nicox Clinical Site, Memphis, Tennessee
  - Nicox Clinical Site, Austin, Texas
  - Nicox Clinical Site, El Paso, Texas
  - Nicox Clinical Site, Houston, Texas
  - Nicox Clinical Site, Mission, Texas
  - Nicox Clinical Site, San Antonio, Texas
  - Nicox Clinical Site, Sugar Land, Texas
  - Nicox Clinical Site, St. George, Utah
  - Nicox Clinical Site, Falls Church, Virginia
  - Nicox Clinical Site, Bellevue, Washington
  - Nicox Clinical Site, Seattle, Washington
- China (20):
  - Nicox Clinical Site, Lanzhou, Gansu
  - Nicox Clinical Site, Shantou, Guangdong
  - Nicox Clinical Site, Harbin, Heilongjiang
  - Nicox Clinical Site, Zhengzhou, Henan
  - Nicox Clinical Site, Wuhan, Hubei
  - Nicox Clinical Site, Yichang, Hubei
  - Nicox Clinical Site, Changsha, Hunan
  - Nicox Clinical Site, Changsha, Huna
  - Nicox Clinical Site, Nanchang, Jiangxi
  - Nicox Clinical Site, Changchun, Jilin
  - Nicox Clinical Site, Dalian, Liaoning
  - Nicox Clinical Site, Xi'an, Shaanxi
  - Nicox Clinical Site, Jinan, Shandong
  - Nicox Clinical Site, Qingdao, Shandong
  - Nicox Clinical Site, Chengdu, Sichuan
  - Nicox Clinical Site, Wenzhou, Xhejiang
  - Nicox Clinical Site, Beijing
  - Nicox Clinical Site, Chongqing
  - Nicox Clinical Site, Shanghai
  - Nicox Clinical Site, Tianjing

IPD SHARING:
Plan to Share IPD: No